CLINICAL TRIAL: NCT05439057
Title: Effect of Remimazolam on Postoperative Nausea and Vomiting in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Effect of Remimazolam on Postoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, In-Jung Jun, associate professor, Inje University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 2022-03-007
Record Dates: First submitted 2022-06-27; First posted 2022-06-30 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — remimazolam; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Remimazolam group (Experimental): Remimazolam is started during induction of anesthesia at the rate of 0.3 mg/kg/hr and stopped 20 minutes before end of operation.
  Interventions: Drug: Remimazolam
- Control group (Placebo Comparator): 0.9% normal saline is started during induction of anesthesia at the rate of 0.3 ml/kg/hr and stopped 20 minutes before end of operation.
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Remimazolam — Remimazolam is infused at a rate of 0.3 mg/kg/hr from induction of anesthesia until 20 minutes before the end of operation.
  Other Names: remimazolam group
  Arms: Remimazolam group
Drug: Control — Normal saline is infused at a rate of 0.3 ml/kg/hr from induction of anesthesia until 20 minutes before the end of operation.
  Other Names: control group
  Arms: Control group

SUMMARY:
The present trial is to study the effect of low dose remimazolam on postoperative nausea and vomiting (PONV) in patients at risks of PONV (women, postoperative use of opioid, nonsmokers) undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is a common complication in patients undergoing general anesthesia. It is reported that PONV is observed in 50% of patients 24 hours after general anesthesia and upto 80% in high risk patients. The patients experiencing PONV may experience severe discomfort that it is important to prevent PONV. There are several prophylactic agents for PONV. 5 serotonin receptor antagonist(5-HT3 antagonist) is the most commonly used agent and other agents such as corticosteroid, neurokinin-1 receptor antagonist can also be used. Previous studies have reported the efficacy of benzodiazepine(midazolam) in a low targeting dose as a prophylactic agent of PONV. The efficacy of low dose remimazolam (short acting benzodiazepine) on PONV has not been evaluated.

According to Fourth consensus guideline for the management of postoperative nausea and vomiting (2020), three prophylactic anti-emetics are recommended for patients with three or more of the risk factors of PONV. As the patients included in our study have three or more of risk factors of PONV (women, postoperative use of opioid, nonsmokers), three prophylactic anti-emetics are recommended. Our center has routinely been using 5-HT3 receptor antagonist (ramosetron) and corticosteroid (dexamethasone) for women undergoing laparoscopic cholecystectomy. However, we still find many patients complaining nausea and vomiting after operation. Therefore, we are willing to investigate the low supplemental dose of remimazolam on the prophylaxis of PONV.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing laparoscopic cholecystectomy under general anesthesia.

Exclusion Criteria:

* moderate to severe liver dysfunction (total bilirubin ≧ 3.0 mg/dL / aspartate aminotransferase(AST) or alanine aminotransferase(ALT) ≧ 2.5 times more than normal range)
* moderate to severe renal dysfunction (serum creatinine ≧ 2.0 mg/dL / end-stage renal disease undergoing hemodialysis)
* tolerance to benzodiazepines
* hypersensitivity to anesthetic drugs (Benzodiazepines, Propofol, Remifentanil, Fentanyl citrate, Rocuronium bromide, Flumazenil)
* acute angle glaucoma
* alcohol dependence
* Galactose intolerance, Lactase deficiency, glucose-galactose malabsorption
* pregnant, breast feeding women
* BMI >35 kg/m2
* uncontrolled diabetes mellitus

Ages: 19 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2022-04-13 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
postoperative nausea and vomit within 24 hours after the end of operation | Upto 24 hours after surgery
  Nausea is evaluated using 11-point verbal numeric rating scale (VNRS -none:0, mild: 1-3, moderate:4-6, severe 7-10). Vomiting is checked when the patient has vomited or has retching symptom.

SECONDARY OUTCOMES:
quality of recovery (QoR-15) 24 hours after the end of the operation | Upto 24 hours after surgery
  QoR-15 survey is performed 24 hours after the end of the operation.
pain 24 hours after the end of the operation | Upto 24 hours after surgery
  pain is evaluated using Numeric rating scale (NRS).

CONTACTS AND LOCATIONS:
Overall Officials: In-Jung Jun, MD.PhD., Principal Investigator — Associate professor
Locations (1):
- Sanggye Paik hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park S, Yon JH, Lee S, Kim KM, Jun IJ. Efficacy of intraoperative low-dose remimazolam as a third antiemetic agent for preventing early postoperative nausea in high-risk patient: A Randomized controlled trial. BMC Anesthesiol. 2025 Sep 2;25(1):442. doi: 10.1186/s12871-025-03332-3. PMID 40898019